CLINICAL TRIAL: NCT06982209
Title: Analgesia/Nociception Index (ANI)-Guided Desflurane Titration Reduces Anesthetic Consumption in Laparoscopic Cholecystectomy: A Prospective Randomized Controlled Trial
Brief Title: ANI-Guided Anesthetic Desflurane Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Cheol Lee,MD,PhD,, Professor, Wonkwang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Wonkwang UH20
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Pain; General Anesthesia; Laparoscopic Cholecystectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Analgesia

STUDY DESIGN:
Intervention Model Description: * ANI Group: Desflurane started at 1 MAC (~6 Vol%), titrated in 0.1 MAC increments to maintain ANI 50-70 and BIS 40-60. ANI <50 prompted an increase; ANI >70 prompted a decrease.
  * Control Group: Desflurane was titrated based on vital signs (heart rate, blood pressure) and BIS 40-60, per institutional protocol.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, care providers (excluding anesthesiologists), and outcome assessors were blinded to group allocation. Anesthesiologists administering anesthesia were unblinded due to the requirement for ANI monitoring and titration in the intervention group. Outcome assessors in the PACU were independent staff blinded to intraoperative management.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ANI-guided group (Experimental): Desflurane started at 1 MAC (~6 Vol%), titrated in 0.1 MAC increments to maintain ANI 50-70 and BIS 40-60. ANI <50 prompted an increase; ANI >70 prompted a decrease
  Interventions: Device: Analgesia/Nociception Index (ANI)
- Control group (Active Comparator): Desflurane was titrated based on vital signs (heart rate, blood pressure) and BIS 40-60, per institutional protocol.
  Interventions: Device: Analgesia/Nociception Index (ANI)

INTERVENTIONS:
Device: Analgesia/Nociception Index (ANI) — ANI was monitored using the ANI monitor (MetroDoloris, France) in both groups, but only guided adjustments in the ANI group

SUMMARY:
General anesthesia requires precise titration of inhaled anesthetics like desflurane and opioids like remifentanil to balance sedation, analgesia, and hemodynamic stability. The Analgesia/Nociception Index (ANI), derived from heart rate variability (HRV), quantifies parasympathetic tone to assess nociception-antinociception balance on a 0-100 scale, with lower values indicating nociceptive stress. ANI analyzes high-frequency HRV components, reflecting parasympathetic inhibition during painful stimuli, making it a reliable indicator of intraoperative nociception. Studies validate the utility of ANI in detecting nociceptive events during laparoscopic surgery. ANI-guided opioid titration reduces opioid consumption and stabilizes hemodynamics, enhancing perioperative outcomes.

DETAILED DESCRIPTION:
Study Design This prospective, single-center, randomized controlled trial receives approval from the [Institutional Review Board Name] (Approval No. 2024-01-05-21-004). Written informed consent is obtained from all participants.

Participants Eligible patients are aged 19-65 years, American Society of Anesthesiologists (ASA) physical status I-II, and are scheduled for elective laparoscopic cholecystectomy under general anesthesia. Exclusion criteria include chronic pain, preoperative opioid use, cardiac arrhythmias, autonomic dysfunction, or contraindications to desflurane or remifentanil.

Randomization and Blinding Patients are randomized (1:1) to Analgesia/Nociception Index (ANI)-guided or standard care groups using a computer-generated sequence in blocks of four. Group allocation is concealed in opaque, sealed envelopes, which are opened before induction. Anesthesiologists remain unblinded due to ANI monitoring requirements, but patients and postoperative outcome assessors remain blinded to reduce bias.

Anesthesia Protocol Anesthesia is induced with propofol (2 mg/kg) and rocuronium (0.6 mg/kg). Maintenance includes desflurane and remifentanil (0.1 µg/kg/min continuous infusion). Ventilation maintains normocapnia (end-tidal Carbon dioxide: 35-40 mmHg). Bispectral index (BIS) is monitored to ensure hypnotic depth (target: 40-60).

Novel Metrics

In addition to standard intraoperative management, the following novel physiological and recovery-related metrics are assessed to enhance the evaluation of ANI-guided anesthesia:

* ∆ANI (Dynamic Change of ANI): The percentage change in ANI at specific surgical stimuli (e.g., skin incision, trocar insertion) is recorded as: ∆ANI = (ANI_post - ANI_pre) / ANI_pre × 100.
* Autonomic Nervous System Indicators:
* Heart Rate Variability (HRV): High Frequency (HF) and Low Frequency (LF)/HF ratio are calculated at baseline, mid-surgery, and end-surgery. Continuous beat-to-beat blood pressure (BP) and lead II electrocardiogram (ECG) are recorded noninvasively for 5 minutes using the equipment. HRV parameters are extracted using Software.
* Baroreflex Sensitivity (BRS): BRS is assessed pre-induction and intraoperatively. It is quantified using the spontaneous sequence method with regression analysis between Blood Pressure and respiratory rate intervals, measured with the equipment and analyzed with HRV Software.

Recovery Room Metrics

* Post-Anesthesia Care Unit (PACU) Length of Stay (LOS): Time from PACU entry to discharge readiness is recorded.
* Additional Analgesic Requirement: Any supplemental pain medication and dosage are recorded during PACU stay.
* Postoperative Nausea and Vomiting (PONV): Incidence is recorded within the first two postoperative hours.

Patient-Reported Outcomes

* Satisfaction Scores (Visual analogue scale [VAS]0-10): Are assessed at PACU discharge and on postoperative day 1 (POD1).
* ANI Group: Desflurane starts at 1 Minimum Alveolar Concentration (MAC) (~6 Vol%) and is titrated in 0.1 MAC increments to maintain ANI 50-70 and BIS 40-60. ANI <50 prompts an increase; ANI >70 prompts a decrease.
* Control Group: Desflurane is titrated based on vital signs and BIS 40-60 per institutional protocol.

ANI is monitored using the ANI monitor in both groups, but only guides adjustments in the ANI group. Hemodynamic data are recorded every 5 minutes.

Emergence and Recovery At the end of the surgery, desflurane and remifentanil are discontinued. Neuromuscular blockade is monitored using Train-of-Four (TOF) stimulation. When TOF count reaches ≥2, sugammadex (2 mg/kg) is administered to reverse rocuronium. Extubation occurs when TOF ratio >0.9, with adequate spontaneous breathing and responsiveness to verbal commands. Emergence time is recorded as time from anesthetic cessation to eye opening.

Outcome Measures

* Primary Outcome: Mean end-tidal desflurane concentration (Vol%).
* Secondary Outcomes:
* Emergence time (min).
* Postoperative pain (VAS, 0-10) at 30 min post-extubation.
* Intraoperative hemodynamic stability (hypertension [Mean arterial pressure > 100 mmHg] or tachycardia [HR >100 bpm]).
* ∆ANI at surgical stimuli.
* HRV metrics (HF, LF/HF ratio).
* Baroreflex Sensitivity (BRS).
* PACU LOS.
* Requirements and dosage of additional analgesics in PACU.
* Incidence of PONV within 2 hours post-op.
* Patient satisfaction (PACU discharge and postoperative day 1).

ELIGIBILITY:
Inclusion Criteria:

* aged 19-65 years, American Society of Anesthesiologists (ASA) physical status I-II, scheduled for elective laparoscopic cholecystectomy under general anesthesia.

Exclusion Criteria:

* chronic pain, preoperative opioid use, cardiac arrhythmias, autonomic dysfunction, or contraindications to desflurane or remifentanil.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Mean End-Tidal Desflurane Concentration | From induction of anesthesia to end of surgery (approximately 60 minutes)
  The average end-tidal desflurane concentration (Vol%) during maintenance of general anesthesia, measured using continuous gas monitoring. Desflurane delivery is titrated based on ANI (Analgesia/Nociception Index) in the intervention group and based on vital signs in the control group.

SECONDARY OUTCOMES:
Emergence Time | At the end of surgery until eye opening (approximately 5-15 minutes)
  Time from discontinuation of anesthetics to eye opening upon verbal command, recorded in minutes.
Post-Anesthesia Care Unit (PACU) Length of Stay | From PACU entry to PACU discharge criteria fulfillment (approximately 30-90 minutes)
  Time from PACU admission to discharge readiness, measured in minutes.
Additional Analgesic Requirement in PACU | During PACU stay (up to 2 hours after surgery)
  Number of patients requiring additional analgesics in PACU and total morphine-equivalent dose administered.
Incidence of Postoperative Nausea and Vomiting (PONV) | Within 2 hours after surgery
  Presence of nausea or vomiting events recorded within the first two postoperative hours.
Patient Satisfaction | At PACU discharge and 24 hours postoperatively (POD1)
  Patient-reported satisfaction using a Visual Analog Scale (0-10) at PACU discharge and on postoperative day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Lee, M.D.,Ph.D, Principal Investigator — Wonkwang University Hospital
Locations (1):
- Wonkwang University School of Medicine Hospital, Iksan, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No